CLINICAL TRIAL: NCT04722419
Title: Factors That Determine the Responses to Meal Ingestion in Functional Dyspepsia
Brief Title: Responses to a Comfort Meal in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016L
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: meal ingestion; postprandial responses; hedonic sensations; homeostatic sensations; functional dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional dyspepsia (Experimental)
  Interventions: Other: Probe meal
- Healthy subjects (Active Comparator)
  Interventions: Other: Probe meal

INTERVENTIONS:
Other: Probe meal — The probe meal will be served in 112 Kcal portions (16 g white bread, 10 g cheese, 10 g jam, 3.25 g butter, and 50 mL orange juice) up to the level of maximal satiation.

SUMMARY:
Background. Dyspeptic patients tolerate smaller meal loads than healthy subjects, but it is not known whether and to what extent symptoms relate to abnormal homeostatic or hedonic components of perception. Methods. Parallel studies in patients with symptoms induced by meals (fulfilling Rome IV criteria of postprandial dyspepsia) and sex- and age-matched healthy subjects. Participants will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 4 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Participants will ingest a probe meal up to the level of maximal satiation. The probe meal will be served stepwise (112 Kcal every 5 min). Perception of homeostatic (hunger/satiation, fullness) and hedonic (digestive well-being, mood) sensations will be measured at 5 min intervals 10 min before, during and 20 min after ingestion at 10 min intervals.

ELIGIBILITY:
Inclusion Criteria for Patients with Functional Dyspepsia:

* Rome IV Criteria for Functional Dyspepsia

Inclusion Criteria for Healthy Subjects

* absence of digestive symptoms

Exclusion Criteria for all participants:

* history of anosmia and ageusia
* alcohol abuse
* psychological disorders
* eating disorders

Inclusion Criteria for Healthy Subjects:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Meal enjoyment | 100 minutes
  Amount of meal (Kcal) consumed up to the level of maximal digestive well-being measured on a - 5 (extremely unpleasant sensation) to + 5 scale (extremely pleasant sensation).

SECONDARY OUTCOMES:
Change in digestive well-being induced by the probe meal | 1 day
  Change in well-being measured by 10 score scales during and after the probe meal.
Change in fullness sensation induced by the probe meal | 1 day
  Change in fullness sensation measured by 10 score scales during and after the probe meal.
Change in mood induced by the probe meal | 1 day
  Change in mood measured by 10 score scales during and after the probe meal.
Change in abdominal discomfort induced by the probe meal | 1 day
  Change in abdominal discomfort measured by 10 score scales during and after the probe meal.
Change in hunger/satiety induced by the probe meal | 1 day
  Change in hunger/satiety measured by 10 score scales during and after the probe meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Livovsky DM, Pribic T, Azpiroz F. Food, Eating, and the Gastrointestinal Tract. Nutrients. 2020 Apr 2;12(4):986. doi: 10.3390/nu12040986. PMID 32252402